CLINICAL TRIAL: NCT04182126
Title: Environmental Modifications in Sub-Saharan Africa: Changing Epidemiology, Transmission and Pathogenesis of Plasmodium Falciparum and P. Vivax Malaria
Brief Title: Adaptive Interventions for Optimizing Malaria Control: a Cluster-Randomized SMART Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Guiyun Yan, Professor, University of California, Irvine
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 20173512
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-05

CONDITIONS: LLIN, PBO LLIN, IRS, Larviciding
Keywords: Adaptive intervention; Multiple assignment randomized trial (SMART); Cluster-randomized SMART trial; Optimal intervention strategy; Clinical malaria incidence; Cost-effectiveness

STUDY DESIGN:
Intervention Model Description: This study will use a longitudinal sequential multiple assignment randomized trial design. It will include multiple stages, at each stage, clusters are assigned to different arms (interventions) using an adaptive strategy. Therefore, number of arms vary from stage to stage.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study partially masking participants, because by design some participants will receive PBO treated long-lasting insecticidal nets (LLINs) and others will not receive such bed nets, therefore, those who receives the PBO LLINs can not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Regular long-lasting insecticidal nets (Placebo Comparator): All participants will have LLIN coverage through routine MoH distribution of long-lasting insecticidal nets (LLINs), no other interventions will be applied. Regular LLIN: Olyset nets containing 2% permethrin or PermaNet 2.0 containing 1.8 and 1.4 g/kg, respectively, for 75 and 100 denier yarn.
  Interventions: Other: Regular long-lasting insecticidal nets
- Piperonyl butoxide-treated LLIN (Experimental): All participants will received piperonyl butoxide-treated LLINs (PBO-LLINs) at Stage 1 and Stage 2 interventions provided that PBO-LLINs are effective at Stage 1 interventions. Each household will be provided on PBO-LLIN per two people with appropriate eduction.
  PBO-LLIN: Olyset Plus, containing 2% permethrin and 1% PBO.
  Interventions: Other: LLIN plus Piperonyl butoxide-treated LLIN
- PBO-LLIN plus larval source management (Experimental): All participants will received piperonyl butoxide-treated LLINs (PBO-LLINs) at Stage 1. However, if Stage 1 intervention is not effective, half of them will randomized to receive PBO-LLINs plus larval source management (LSM) at Stage 2. LSM will be implemented in selected clusters, including chemical methods by larviciding of semi-permanent and permanent habitats, per the National Malaria Strategic Plan of Kenya. The investigators will use the long-lasting microbial larvicides manufactured by Central Life Sciences. Semi-permanent and permanent habitats will be treated with FourStar® 180-day Briquets using the recommended dosage of 100 ft2 water surface per briquet.
  Interventions: Other: LLIN plus Piperonyl butoxide-treated LLIN; Other: Long-lasting microbial larvicide
- PBO-LLIN plus enhanced methods (Experimental): All participants will received piperonyl butoxide-treated LLINs (PBO-LLINs) at Stage 1, however, Stage 1 intervention is not effective. All participants will received PBO-LLINs plus an enhanced intervention at Stage 2, i.e., annual IRS using Kenya Government recommended insecticides.
  Interventions: Other: LLIN plus Piperonyl butoxide-treated LLIN
- LLIN plus indoor residual spraying (Experimental): All participants will received regular LLINs plus indoor residual spraying (IRS) (LLIN+IRS) at Stage 1 and Stage 2 interventions provided that LLIN+IRS is effective at Stage 1 interventions. For LLIN+IRS clusters, each dwelling's interior walls and ceilings will be sprayed with micro-encapsulated pirimiphos-methyl (Actellic 300CS) at the recommended dosage of 1g/m² and at the government-recommended frequency. If Kenya government switch the IRS insecticide, the investigators will use the same insecticide as the government recommended.
  Interventions: Other: Regular long-lasting insecticidal nets; Other: Indoor residual spraying with micro-encapsulated pirimiphos-methyl or other insecticides
- LLIN+IRS twice a year (Experimental): All participants will received regular LLINs plus IRS at Stage 1, provided that LLIN+IRS is not effective. IRS will be increased to twice a year.
  Interventions: Other: Regular long-lasting insecticidal nets; Other: Long-lasting microbial larvicide; Other: Indoor residual spraying with micro-encapsulated pirimiphos-methyl or other insecticides
- LLIN+IRS plus enhanced method (Experimental): All participants will received regular LLINs plus IRS at Stage 1, provided that LLIN+IRS is not effective. Enhanced method will be added on these clusters at Stage 2 interventions.The enhanced intervention is the regular IRS plus IRS treating animal sheds and other outdoor structures.
  Interventions: Other: Regular long-lasting insecticidal nets; Other: Indoor residual spraying with micro-encapsulated pirimiphos-methyl or other insecticides

INTERVENTIONS:
Other: Regular long-lasting insecticidal nets — Olyset nets: containing 2% permethrin or PermaNet 2.0 containing 1.8 and 1.4 g/kg, respectively, for 75 and 100 denier yarn
  Other Names: LLIN
  Arms: LLIN plus indoor residual spraying; LLIN+IRS plus enhanced method; LLIN+IRS twice a year; Regular long-lasting insecticidal nets
Other: LLIN plus Piperonyl butoxide-treated LLIN — Olyset Plus: containing 2% permethrin and 1% PBO
  Other Names: PBO-LLIN
  Arms: PBO-LLIN plus enhanced methods; PBO-LLIN plus larval source management; Piperonyl butoxide-treated LLIN
Other: Long-lasting microbial larvicide — Semi-permanent and permanent habitats will be treated with FourStar® 180-day Briquets using the recommended dosage of 100 ft2 water surface per briquet
  Other Names: FourStar® 180-day Briquets
  Arms: LLIN+IRS twice a year; PBO-LLIN plus larval source management
Other: Indoor residual spraying with micro-encapsulated pirimiphos-methyl or other insecticides — Each dwelling's interior walls and ceilings will be sprayed with micro-encapsulated pirimiphos-methyl at the recommended dosage of 1g/m² and at the recommended frequency of once a year or twice a year. Other insecticides may be used to replace the Actellic 300 CS depends on Kenya government policy, current policy requires rotating different insecticides annually.
  Other Names: Actellic 300CS or Kenya government recommended insecticdes
  Arms: LLIN plus indoor residual spraying; LLIN+IRS plus enhanced method; LLIN+IRS twice a year

SUMMARY:
In the past decade, massive scale-up of long-lasting insecticidal nets (LLINs) and indoor residual spraying (IRS) have led to significant reductions in malaria mortality and morbidity. Nonetheless, malaria burden remains high, and a dozen countries in Africa show a trend of increasing malaria incidence over the past several years. The high malaria burden in many areas of Africa underscores the need to improve the effectiveness of intervention tools by optimizing first-line intervention tools and integrating newly approved products into control programs. Vector control is an important component of the national malaria control strategy in Africa. Because transmission settings and vector ecology vary among countries or among districts within a country, interventions that work in one setting may not work well in all settings. Malaria interventions should be adapted and re-adapted over time in response to evolving malaria risks and changing vector ecology and behavior. The central objective of this application is to design optimal adaptive combinations of vector control interventions to maximize reductions in malaria burden based on local malaria transmission risks, changing vector ecology, and available mix of interventions approved by the Ministry of Health in each target country. The central hypothesis is that an adaptive approach based on local malaria risk and changing vector ecology will lead to significant reductions in malaria incidence and transmission risk. The aim of this study is to use a cluster-randomized sequential, multiple assignment randomized trial (SMART) design to compare various vector control methods implemented by the Ministry of Health of Kenya in reducing malaria incidence and infection, and develop an optimal intervention strategy tailored toward to local epidemiological and vector conditions.

DETAILED DESCRIPTION:
In the past decade, massive scale-up of long-lasting insecticide-treated nets (LLINs) and indoor residual spraying (IRS) in Africa have led to significant reductions in malaria mortality and mobility. However, current first-line interventions are not sufficient to eliminate malaria in most countries. The widespread use of pyrethroid insecticides has resulted in resistant vector populations, and high coverage of LLINs and IRS has led to increased outdoor human feeding behavior and resting behavior. These changes in vector ecology and behaviors have significantly limited the effectiveness of current first-line interventions that target indoor biting and resting mosquitoes. Furthermore, as a result of ecological changes and intervention measures, malaria risk in a locality is dynamic, and the utility of malaria intervention tools may vary as new tools are being approved and introduced and the cost of each tool differs among locations and over time. Such variations in malaria risk, vector ecology, and utility of intervention tools exemplify the need to develop optimal adaptive interventions tailored to local malaria risks, vector ecology and supply chains. The central objective of this application is to design optimal adaptive combinations of vector control interventions to maximize reductions in malaria burden based on local malaria transmission risks, changing vector ecology, and available mix of interventions approved by the Ministry of Health in each target country. The central hypothesis is that an adaptive approach based on local malaria risk and changing vector ecology will lead to significant reductions in malaria incidence and transmission risk. To accomplish this objective, the investigators propose the following three specific aims:

1. Measure malaria incidence and predict risk using environmental, biological, social, and climatic features with machine learning approaches. Hypothesis: Malaria risk prediction can be improved through the use of machine learning techniques that include environmental, biological, socioeconomic, and climatic features. Approach: Each site will measure malaria incidence, prevalence and social economic factors through community surveys. Classification-based and regression-based approaches will be used to develop malaria risk predictive models, and model performance will be validated. Outcome: This Aim will establish improved malaria risk prediction models and lay an important foundation for developing intervention strategies adaptive to local vector ecology and future malaria risks using reinforced machine learning approaches.
2. Use a cluster-randomized sequential, multiple assignment randomized trial (SMART) design to develop an optimal adaptive intervention strategy. Hypothesis: Malaria control interventions that are adapted to local malaria risk and vector ecology and are cost effective can be identified using a cluster-randomized SMART design. Approach: Cluster-randomized SMART design will be used in a high transmission areas in Kenya to evaluate the impact of adaptive interventions that involve sequential and combination use of next-generation nets, indoor spraying of non-pyrethroid insecticides, and larval source management for malaria control.
3. Evaluate the cost-effectiveness and impact of an adaptive intervention approach on secondary endpoints related to malaria risk and transmission. Hypothesis: Intervention strategies adapted to local malaria risk and vector ecology will be more cost-effective in reducing malaria incidence and transmission risk than the currently-used LLIN intervention. Approach: The economic costs of individual interventions or combinations thereof will be assessed from both a provider and societal perspective using standard economic evaluation methodologies. Cost-effectiveness will be measured in terms of cost per person protected. The study will examine changes in drug and insecticide resistance and infection prevalence attributable to the adaptive interventions.

Malaria interventions adapted to rapidly changing malaria risk and vector ecologies are critically needed to improve the effectiveness of malaria control measures. This study will use new techniques, including machine learning and a novel cluster-randomized SMART design, to develop optimal adaptive malaria intervention strategies.

The investigators will use 84 clusters in Kisumu County in Western Kenya to conduct the trial. Since it is a sequential multiple assignment randomized trail, the trial will include several intervention stages. At each stage there will be different interventions. If an intervention is effective (i.e., yields an above threshold reduction in malaria incidence) at Stage 1, the intervention will be continued, otherwise, the intervention will be replaced by another one at Stage 2. The replacement intervention may be decided by different ways, e.g., an known effective intervention or an intervention determined by a machine learning algorithm. Since interventions in some clusters may be continued (i.e., effective) by next stage, other interventions may be replaced by different interventions, the number of interventions arms can vary from stage to stage. This is very different from ordinary cluster randomized trials. In this trial, the investigators planned to start with piperonyl butoxide (PBO) treated long-lasting insecticidal nets (PBO LLIN), indoor residual spraying with Actellic(R) insecticide, and using the routine LLIN intervention as control. Both Actellic IRS and PBO LLIN have been tested to be effective against pyrethroid resistant Anopheles malaria vectors and reduce clinical malaria. Therefore, the initial stage will have three arms, i.e., regular LLIN, PBO LLIN, and regular LLIN plus Actellic IRS. Since the investigators don't know if the effectiveness of these interventions in different clusters, the stage 2 interventions may include up to 7 arms, i.e., some arms may be split into two arms, based on the evaluation at the end of Stage 1 intervention.

The investigators will begin the trial with a two-year smaller scale trial using 36 cluster and randomly assign the three interventions, i.e., regular LLIN, PBO LLIN and regular LLIN plus Actellic IRS, into these 36 cluster, with 12 clusters for each intervention. This pre-trial trial is to determine the optimal way for conducting the full-scale 84 cluster trial, including operational and effectiveness evaluation procedures, as well as cost-effectiveness analysis. The full scale 84 cluster trial will be started by Year 3. The full trial will be started from fresh, i.e., the same three interventions will be randomly assigned to the 84 clusters with 28 clusters for each interventions. Clinical malaria will be monitored using a cohort active case surveillance, parasite prevalence and vector density will be monitored using cross-sectional samplings. The results of these surveillance at the end of Stage 1 trial will be used to evaluate the effectiveness of interventions at each cluster for the Stage 1 interventions. Stage 2 interventions will be determined for each cluster based on the above evaluations, e.g., continue the same intervention or replace the intervention with different ones.

ELIGIBILITY:
Household inclusion criteria:

* Households with residents at the time of survey
* Agreement of the adult resident to provide informed consent for the intervention and survey

Study subjects inclusion criteria:

* Passive case detection by health facilities will include all residents in the study clusters; active case detection will include residents of >6 months
* Agreement of parent/guardian to provide informed consent and minors to provide assent.

Household exclusion criteria:

* Household vacant
* No adult resident home on more than 3 occasions

Study subjects exclusion criteria:

• Participants not home on day of survey

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122872 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Annual clinical malaria incidence rate | Clinical malaria will be monitored for up to 60 months
  To compare clinical malaria incidence rates among different intervention arms

SECONDARY OUTCOMES:
Malaria infection prevalence | Infection prevalence will be monitored for up to 60 months
  To compare infection prevalence rates among different intervention arms using microscopic, RDT and molecular diagnostic methods
Malaria vector density | Vector density will be monitored for up to 60 months
  To compare malaria vector densities between different intervention arms
Malaria transmission intensity | Entomological inoculation rate will be examined for up to 60 months
  To compare entomological inoculation rates between different intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Guiyun Yan, Ph.D., Principal Investigator — University of California at Irvine; John Githure, Ph.D., Study Director — Tom-Mboya University, Kenya
Locations (2):
- Program in Public Health, Irvine, California, United States
- Tom-Mboya University College, Maseno University, Homa Bay, Homa Bay County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou G, Lee MC, Atieli HE, Githure JI, Githeko AK, Kazura JW, Yan G. Adaptive interventions for optimizing malaria control: an implementation study protocol for a block-cluster randomized, sequential multiple assignment trial. Trials. 2020 Jul 20;21(1):665. doi: 10.1186/s13063-020-04573-y. PMID 32690063